CLINICAL TRIAL: NCT01492907
Title: Pilot Study of Meat-Borne Carcinogens and Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011NTLS016
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Pancreatic Cancer
Keywords: Heterocyclic amine carcinogens; meat-borne carcinogens
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Control Participants (Active Comparator): age/sex matched normal controls - the subject will swallow a capsule with a dietary relevant dose of MeIQx
  Interventions: Radiation: MeIQx
- Pancreatic Cancer Patients (Active Comparator): Patients with operable pancreatic cancer scheduled for a pancreatectomy at the University of Minnesota Medical Center.
  Interventions: Radiation: MeIQx; Procedure: Pancreatectomy

INTERVENTIONS:
Radiation: MeIQx — On the day of administration, the subject will swallow a capsule with a dietary relevant dose of MeIQx, 21 µg, labeled with a very low level of 14-carbon. The radioactive dose for MeIQx, 0.002 mSv (4.3 µCi), or less than an average dental x-ray.
  Other Names: [14C]-MeIQx (2 Amino-3,8-dimethylimidazo[4,5 f]quinoxaline-2-[14C])
Procedure: Pancreatectomy — Patients with operable pancreatic cancer scheduled for a pancreatectomy at the University of Minnesota Medical Center.
  Arms: Pancreatic Cancer Patients

SUMMARY:
Study Design:

This is a single institution pilot study to recruit 4 patients with operable pancreatic cancer scheduled for a pancreatectomy and 4 age/sex matched normal controls. Both groups will receive a single oral dose of radiolabeled MelQx followed by serial blood draws over an 8 hour period and urine collections over a 24 hour period. In addition, normal pancreatic tissue and normal small bowel tissue will be collected by Tissue Procurement from resected (waste) tissue at the time of pancreatectomy on the 4 pancreatic cancer patients.

DETAILED DESCRIPTION:
This is not a therapeutic trial. It is an etiologic investigation of meat-borne carcinogens and possible role in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

Cancer cases are eligible for participation if all of the following criteria are met:

* 1. Diagnosis or suspected diagnosis of pancreatic or periampullary cancer that is deemed to be operable and for which a pancreatectomy is planned.
* At least 18 years of age.
* Adequate hepatic function within 4 weeks of study enrollment defined as:

  * Bilirubin ≤ 2 mg/dl
  * aspartate aminotransferase (ALT), alanine aminotransferase (AST), alkaline phosphatase ≤ 2 the upper limit of normal (ULN)
* Females of childbearing potential or males whose partners are of child bearing potential are required to use an effective method of contraception (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 2 weeks after MelQx administration.
* Voluntary written consent before performance of any study-related procedure not part of normal medical care

Healthy controls are eligible for participation if all of the following criteria are met:

* Consider themselves generally healthy.
* At least 18 years of age
* Controls will be gender and age matched within 10 years of cases.
* Adequate hepatic function within 4 weeks of study enrollment defined as:

  * Bilirubin ≤ 2 mg/dl
  * ALT, AST, alkaline phosphatase ≤ 2 the upper limit of normal (ULN)
* Females of childbearing potential or males whose partners are of child bearing potential are required to use an effective method of contraception (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 2 weeks after MelQx administration.
* Voluntary written consent before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

Cancer cases are not eligible for participation if any of the following criteria are met:

For the purposes of this study to reduce the risk of recruiting a potentially unresectable patient:

* Tumor ≥ 3 cm by scan
* CA-19-9 > 400
* Ascites
* Pregnant or lactating
* Uncontrolled chronic conditions such as: cardiovascular disease, hypertension, angina, congestive obstructive pulmonary disease (COPD) or other conditions which may alter metabolism, other than diabetes.

Healthy controls are not eligible for participation if any of the following criteria are met:

* Pregnant or lactating.
* Uncontrolled chronic conditions such as cardiovascular disease, hypertension, angina, COPD or conditions which may alter metabolism including diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Metabolite Profile of Radiolabeled MeIQx in Blood | Pre MeIQx Administration, 1/2, 1, 2, 4, 6, 8 Hours Post MeIQx Administration
  Metabolite levels will be expressed as the percent of total recovered radioactivity in plasma. Metabolite profiles will be qualitatively compared between cases and controls, which will include the mean, median, standard deviation, range and 90% confidence interval for the major detoxification metabolites.
Pharmacokinetic Metabolite Profile of Radiolabeled MeIQx in Urine | 0-4, 4-8 and 8-24 Hours Post MeIQx Administration
  Metabolite levels will be expressed as the percent of total recovered radioactivity in urine. Metabolite profiles will be qualitatively compared between cases and controls, which will include the mean, median, standard deviation, range and 90% confidence interval for the major detoxification metabolites.

SECONDARY OUTCOMES:
Quantify [14C]MeIQx-DNA adducts in human pancreas | 4-8 Hours Post MeIQx Administration
  In the pancreatic cancer patients, uninvolved/normal resected (waste) tissue from the surgery will be sent to Lawrence Livermore National Laboratory (LLNL) for DNA extraction following previously published methods. New [14C]MeIQx-DNA adducts formed at physiological concentrations will be detected and quantified in resected tissue with highly sensitive accelerator mass spectrometry (AMS).
Quantify ambient adducts in the human pancreas | 4-8 Hours Post Administration
  DNA adducts already present in resected tissue will be quantified and characterized with a newly improved technique, electrospray capillary high performance liquid chromatography-tandem mass spectrometry (LC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin E. Anderson, Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States